CLINICAL TRIAL: NCT06370221
Title: The Effect of Psoriatic Arthritis on Female Sexual Dysfunction and Their Relation to Sex Hormones
Brief Title: The Effect of Psoriatic Arthritis on Female Sexual Dysfunction
Status: Not yet recruiting | Type: Observational
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Other Study IDs: psoriatic Arthritis
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Cases Group: About 100 patient females suffering from Psoriatic arthritis and to investigate the correlation between sex hormones profile ( estrogen and progesterone level) and female sexual function in Psoriatic arthritis patients
  Interventions: Behavioral: The effect of psoriatic Arthritis
- Group B: Control Group: About 80 healthy control females
  Interventions: Behavioral: The effect of psoriatic Arthritis

INTERVENTIONS:
Behavioral: The effect of psoriatic Arthritis — to assess the frequency rates of sexual problems and associated factors in a cohort of married females with Psoriatic arthritis, and to investigate the correlation between sex hormones profile ( estrogen and progesterone level) and female sexual function in Psoriatic arthritis patients.
  Other Names: Female Sexual dysfunction

SUMMARY:
Psoriasis is one of the most common immunemediated chronic inflammatory skin disorders.

DETAILED DESCRIPTION:
Psoriasis is one of the most common immunemediated chronic inflammatory skin disorders.

Beside genetic factors, several environmental factors such as injuries, infections, stress, drugs, and immune defect take part in autoimmune pathogenesis of the disease. In addition, it has been reported that some hormones may also have a role in the pathogenesis of psoriasis, due to their effects on keratinocytes proliferation.

Studies revealed that sex hormones manifest a variety of biological and immunological effects in the skin which modulate the natural course of psoriasis.

Approximately 20-30% of patients with psoriasis may also have psoriatic arthritis, which often causes significant musculoskeletal pain that significantly impairs quality of life (QoL).

Although sexual dysfunction is a common complaint, affecting 30 to 70% of psoriasis patients, few studies have analyzed the impact of psoriasis and psoriatic arthritis on quality of sexual life.

ELIGIBILITY:
Inclusion Criteria:

* The study will focuses on the relationship between the FSD and PsA;
* The healthy controls will derive from a population within the same geographic area and ethnic background as PsA;
* Used the same questionnaires/instruments of FSFI to diagnose FSD

Exclusion Criteria:

* pregnancy,
* breastfeeding
* being sexually inactive
* having a partner with sexual dysfunction,
* refusing to participate, or
* being unable to read
* Females with any sexual transmitted disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The female sexual function index (FSFI) is a self-reported questionnaire that has been validated in Arabic, and is used to measure a woman's sexual function over the course of the past four weeks.
  A reliable and accurate way to assess female sexual function is the FSFI. The six domains of sexual function-desire, arousal, lubrication, orgasm, satisfaction, and pain-are assessed by the 19 questions in this questionnaire. The response is scored between 0 and 5 on a 5-point Likert scale.
  Disease Activity in Psoriatic Arthritis (DAPSA) Helps measure disease activity in psoriatic arthritis based on joint symptoms, CRP and pain evaluation
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of female sexual function | 6 months
  To identify and understand the mechanisms of sexual problems in Psoriatic arthritis Patients in Qena university hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Qena Hospital, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Undecided